CLINICAL TRIAL: NCT01934426
Title: Identification of Admission High Risk Elderly From Multiple Cohorts: a Pilot Study
Brief Title: Identification of Admission High Risk Elderly
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201303058RINC
Record Dates: First submitted 2013-08-26; First posted 2013-09-04 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Pneumonia; Urinary Tract Infection; Stroke
Keywords: Admission High Risk Elderly
MeSH Terms: conditions — Pneumonia; Urinary Tract Infections; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Admission High Risk: Admission High Risk

SUMMARY:
Objective: The study aim to establish high risk admission model and readmission model for elderly in Taiwan.

Method: Investigators compare the clinical, epidemiological, and socioeconomic characteristics of admitted patients during 1 August,2011 to 31 July,2012. All patients will follow up to end of study to identify 14 days readmission and 30 days readmission to geriatic ward.

Expected Outcomes: (1) To compare the prediction value of derivation cohort and validation cohort. (2) To identify high risk indicators of admission and readmission for elderly. (3) To determine the risk factors in admission elderly association with quality indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age 65 year old above
2. Patients admission to geriatric ward

Exclusion Criteria:

1. Patients with unstable vital sign
2. Patients or dependants reject to sign inform consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study populations include as below; A.Retrospective cohort group B.Perspective cohort group
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Determine percentages of high risk in elderly 14 days readmission to geriatric ward | 1-year
  Readmission in 14 days to geriatric ward is an important issue of elderly.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan